CLINICAL TRIAL: NCT02004223
Title: Phase I Dose Escalation Study of Stereotactic BOOST for Prostate cancER
Brief Title: Early Investigation of High Precision Radiotherapy Prior to Commencing Standard Radiotherapy for Prostate Cancer
Acronym: BOOSTER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal North Shore Hospital (Other)
Responsible Party: Principal Investigator, Professor Thomas Eade, Senior Staff Specialist (Radiation Oncology), Royal North Shore Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13-NSCCRO-P001
Record Dates: First submitted 2013-11-25; First posted 2013-12-09 (Estimated); Last update posted 2021-06-15 (Actual); Status verified 2021-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Dose escalation; Stereotactic; SBRT; Hypofractionation
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dose escalation using stereotactic boost (Experimental): Dose level allocation - Participants will be allocated to the current dose level, or if the current dose level has been filled and acceptable toxicity has been established, they will be enrolled into the next dose level
  Interventions: Radiation: Dose escalation using stereotactic boost

INTERVENTIONS:
Radiation: Dose escalation using stereotactic boost — This is a dose escalation study. Participants will be allocated to the current dose level, or if the current dose level has been filled and acceptable toxicity has been established, they will be enrolled into the next dose level.
  The first dose level will be 20Gy in 2 fractions to PTV and 25Gy to Gross Target Volume (GTV) if identified. The second dose level will be 22Gy in 2 fractions to PTV and 27.5Gy to GTV if identified. The dose level will be 24 Gy in 2 fractions to PTV and 30Gy to GTV if identified.
  Following stereotactic boost, all participants will receive 46Gy in 23 fractions radiotherapy to the prostate / seminal vesicles +/- lymph nodes.

SUMMARY:
Current standard treatment for prostate cancer involves giving patients approximately 40 doses of radiotherapy, one dose per day over an 8 week period. The purpose of this study is to assess the effects of giving two separate high doses of a special type of precision radiotherapy to the prostate and then 5 weeks (instead of 8 weeks) of standard radiotherapy.

Hypothesis: It is safe to give patients an extra two doses of high-precision radiotherapy prior to commencing a shorter period of standard radiotherapy for prostate cancer.

DETAILED DESCRIPTION:
Prostate cancer accounts for one third of all new cancer diagnoses in men and approximately 30% of men will have External Beam Radiotherapy (EBRT) as primary local therapy. Local persistence of prostate cancer treated with radiotherapy is under-appreciated. Prostate cancer has a long natural history and the consequences of local persistence may not be realized for many years.

Prostate cancer has a slow growth with a potential doubling time ranging from weeks to months (median 42 days) which has led to the hypothesis that prostate cancer will behave more like a late reacting tissue(1). Brenner et al. (2) used data from prostate Low Dose Rate (LDR) permanent seed implants and EBRT series to derive an alpha/beta of approximately 1.5. Many groups have also calculated the alpha/beta ratio to be in the < 3.0 range(3).

If the alpha/beta ratio for prostate cancer is lower than the surrounding normal tissues (Brenner et al. have estimated the alpha/beta for the rectum to be over 5.0), doses greater than 2 Gy (hypofractionation) will afford an advantage as there will be a greater sensitivity of prostate cancer to radiation, as compared to the bladder or rectum. This benefit has been exploited for many years with High Dose Rate (HDR) brachytherapy using Iridium -192. Typical doses for HDR are 19Gy in two fractions in addition to 46Gy in 23 fractions of EBRT (4). With reference to our own institutional data from HDR brachytherapy we calculated the dose distribution in recently treated patients. Due to the nature of the iridium dose distribution, there are considerable areas of much higher dose delivered; 200% of the dose (38Gy) to 12.7% of the target volume, 150% (13.75Gy) to 32.6% of the target volume and 125% (11.9Gy) to 60.1% of the target. Despite the high doses to the periphery of the prostate it is possible to limit the dose to the rectum and bladder to 1cc < 75% (14.25Gy) and the 1cc urethra to <125% (23.75Gy) (4). HDR brachytherapy series have reported durable long term Biochemical Failure Free Survival (BFFS), which are as good or better than comparable external beam or surgical series(5). However despite the low toxicity and excellent biochemical outcomes, HDR brachytherapy utilization in Australia is low, with under 300 cases in total per year. This is due to the logistical difficulty of HDR brachytherapy, anaesthetic requirements, nursing care and patient discomfort.

There have been five published studies investigating stereotactic boost in addition to standard fractionation EBRT without using brachytherapy, four reports with the Cyberknife platform (6-9) and one with Intensity Modulated Radiotherapy (IMRT) (10). All of these series have early follow up (FU) with reported BFFS between 77% and 100%. The largest experience is from Katz et al. (8) who reported 73 patients with both intermediate (n= 41) and high risk (n=32) disease. They treated patients with the Cyberknife platform to deliver between 18 and 21 Gy in three fractions in addition to 45 Gy in 25 fractions EBRT. With a median follow up of 33 months, BFFS was 89.5% and 77.7% for the intermediate and high risk patients respectively. A 5 mm expansion from the prostate to the Planned Treatment Volume (PTV) was used except posteriorly, where the margin was 3mm. There was 7% Grade 2 acute genitourinary (GU) and gastrointestinal (GI) toxicity, with late Grade 2 estimates at three years of 5.5% (GU) and 8.2% (GI). Three other series using Cyberknife to mimic HDR were reported between 2008 and 2012 (6, 7, 9). These studies used margins of 0-2 mm posteriorly and 3-5 mm in other directions and reported low rates of Grade 2 and Grade 3 toxicity. Two of these reports specifically attempted to reproduce the heterogeneity of HDR with large areas of the PTV receiving >125% (40% to 45%) and >150% (5% to 10%) of the prescribed dose. Miralbell et al. (10) reported a Linac based IMRT boost in 50 patients in 2010. This series used an endorectal balloon but no image guidance, which may be the cause of their unacceptably high five year estimates of late GI Grade 2 toxicity of 26%.

Primary objective:

The primary study goal is to assess the acute toxicity of Stereotactic Body Radiotherapy (SBRT) boost with three increasing dose levels.

Secondary objectives:

* Nadir PSA at three months and over duration of follow-up
* Three year and five year Freedom From Biochemical Failure (FFBF) (Nadir + 2.0)
* Planning feasibility (Minor and Major planning violations)
* Late Gastrointestinal and Genitourinary Toxicity (modified Radiation Therapy Oncology Group (RTOG) scale)
* Patient reported QOL (EPIC-SF-12)

Hypothesis: It is safe to dose escalate prostate cancer treatment with a stereotactic boost of up to 30Gy in two fractions to the dominant nodule combined with external beam radiotherapy of 46Gy in 23 fractions with < 15% Grade 2 acute morbidity and < 5% Grade 3 acute morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven prostate adenocarcinoma
* PSA obtained within three months prior to enrollment.
* International Prostate Symptom Score (I-PSS) score <15
* No contraindication to MRI (pacemaker, severe claustrophobia)
* Patient must be able to have fiducial markers placed in the prostate (if on anticoagulants, must be cleared by LMO or cardiologist).
* ECOG performance status 0-2
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Previous pelvic radiotherapy
* Prior total prostatectomy
* Unwilling or unable to give informed consent
* Unwilling or unable to complete quality of life questionnaires.

Ages: 35 Years to 85 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2014-01 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | Assessed up to 12 weeks post treatment.
  Portion of patients with grade 3 or greater genitourinary or gastrointestinal toxicity assessed using the Modified Radiation Therapy Oncology Group (RTOG) Toxicity Scale.

SECONDARY OUTCOMES:
Late toxicity | Up to five years
  At a median follow up of 18 months, Kaplan Meir statistics will be used to estimate the 2 year late Gastrointestinal and Genitourinary Toxicity using the modified RTOG scale.
Cumulative toxicity rate: | From the date of treatment completion assessed up to 5 years
  The cumulative incidence of treatment related Grade 2 or higher GI or GU toxicity allowing for competing risk (death without prior toxicity event) and loss to follow up (censoring).
Biochemical failure (PSA failure) | Up to 5 years.
  Nadir PSA at three months and over duration of follow-up. This will be compared to historical controls from our prospective database stratified by initial PSA and androgen deprivation use / duration (nil vs. short term vs. long term).
  When patients have reached a median follow-up of 24 months and 48 months, actuarial Kaplan Meir statistics will be used to estimate the 3 year and 5 year freedom from biochemical failure (FFBF) using the Nadir + 2.0 definition.
change in Quality of Life | From baseline assessed up to 5 years.
  Patient reported QOL using the validated EPIC SF-36 questionnaire will be collected at baseline, 3 months, 9 months and 21-24 months. Analysis will be performed (a) using the mean scores, with a 10 point deterioration deemed clinically significant and (b) as a change from baseline per individual patient using the 21-24 month questionnaire. A 10-20 point deterioration will be deemed mild-moderate and a >20 point deterioration will be deemed significant. Kaplan Meir statistics will be used to estimate the proportion of patients with a ≥10 point, or ≥20 point deterioration at appropriate time points.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas N Eade, MBBS, Principal Investigator — Royal North Shore Hospital
Locations (1):
- Northern Sydney Cancer Centre, Royal North Shore Hospital, St Leonards, New South Wales, Australia